CLINICAL TRIAL: NCT04972695
Title: Validation of an Automatic Analysis Algorithm of the Probability of Glaucoma From Optic Disc Images
Status: Completed | Type: Observational
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Other Study IDs: PI 21-2278
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Glaucoma, Suspect; Glaucoma; Ocular Hypertension
Keywords: Deep Learning; Diagnoses Disease; Glaucoma; retinographies
MeSH Terms: conditions — Ocular Hypertension; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Glaucoma: People with diagnosis of Primary Open Angle Glaucoma (POAG)
  Interventions: Diagnostic Test: Fundus Photographs (retinographies)
- Ocular Hypertension / glaucoma suspect: People with diagnosis of Ocular Hypertension or POAG suspicion
  Interventions: Diagnostic Test: Fundus Photographs (retinographies)

INTERVENTIONS:
Diagnostic Test: Fundus Photographs (retinographies) — Fundus photographs under mydriasis

SUMMARY:
Clinical, cross-sectional and prospective study to assess the images of the posterior pole of the retina of patients from the Glaucoma Unit of the IOBA and the Hospital Clínico Universitario de Valladolid during the period between May and December 2021.

The aim of the project is to provide a sufficient number of images from posterior pole retinographies in patients with suspected glaucoma or with diagnosis of glaucoma in order to determine the sensitivity and specificity of an automatic glaucoma screening algorithm developed by the company Transmural Biotech S.L.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or ocular hypertension
* Signed informed consent
* Visual field examination within the last 12 months

Exclusion Criteria:

* Ocular or systemic pathologies that may interfere with the quality of the retinographic image or the results of the visual field
* Congenital anomalies of the papilla that seriously alter its structure
* High ametropia (> 10 diopters)
* Pharmacological Mydriasis contraindication.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ocular hypertensive patients or patients with diagnosis of Glaucoma.
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of an automated classification system for retinographies | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA - Universidad de Valladolid, Valladolid, Spain